CLINICAL TRIAL: NCT05167292
Title: Acute Kidney Injury Among Adults in the Pacific Islands: Incidence, Aetiology, Management and Outcome Measures From the Tertiary Referral Hospital of Samoa.
Brief Title: Aetiology, Management and Outcomes of Acute Kidney Injury in Samoa.
Status: Completed | Type: Observational
Sponsor: Dr Annette Kaspar (Other Government)
Collaborators: Fiji National University (Other)
Responsible Party: Sponsor-Investigator, Dr Annette Kaspar, Head of Audiology, Tupua Tamasese Meaole Hospital
Organization: Tupua Tamasese Meaole Hospital (Other Government)
Other Study IDs: 117.19
Record Dates: First submitted 2021-11-23; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Acute Kidney Injury
Keywords: Pacific Islands; Incidence; Aetiology; Prevention; Complications
MeSH Terms: conditions — Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Routine clinical care was provided to all AKI cases presenting to the TTM Hospital in Samoa. This prospective observational study reviewed incidence, aetiology and outcomes for these cases.

SUMMARY:
Single-centre prospective observational study. Participants were recruited from the hospital patient information system. The inclusion criteria for participation was (1) adults (>18 years) admitted to general wards of Tupua Tamasese Meaole (TTM) Hospital with a diagnosis of AKI between the 1st December 2019 and the 31st of May 2020, and (2) serum creatinine level of >200 micromol/L, and (3) compliance with the current Kidney Disease Improving Global Outcomes (KDIGO) criteria for AKI diagnosis. The data collection form was adapted from the International Society for Nephrology - Global Snapshot Project, and recorded demographic and baseline characteristics, precipitating causes of AKI, treatment/management, and outcomes measures.

DETAILED DESCRIPTION:
2. METHODS 2.1. Ethical approval Ethical approval for the present study was obtained from the Fiji National University College Health Research Ethics Committee (CHREC) and the Government of Samoa Ministry of Health - Health Research Committee (MoH-HRC). Gatekeeper approval was also obtained from the Deputy Director General of the TTM Hospital.

2.2. Study Design and Data Collection This was a single-centre prospective observational study. Participants were recruited from the hospital patient information system. The inclusion criteria for participation were (1) adults (>18 years) admitted to general wards of Tupua Tamasese Meaole (TTM) Hospital with a diagnosis of AKI between the 1st December 2019 and the 31st of May 2020, and (2) serum creatinine level of >200 micromol/L, and (3) compliance with the current Kidney Disease Improving Global Outcomes (KDIGO) criteria for AKI diagnosis. Patients with underlying chronic kidney disease who experienced an episode of AKI during the study period were also included in the present study. Exclusion criteria were (1) patients on chronic haemodialysis, (2) patients with underlying chronic kidney disease with no evidence of AKI, and (3) patients for whom it was not possible to ascertain a diagnosis (i.e., patients with one elevated serum creatinine result and no subsequent follow-up haematology).

The hospital Laboratory Database was accessed to identify all patients admitted to TTM Hospital during the study period with a serum creatinine level greater than 200 micromol/L. This is higher than the reference intervals for normal creatinine levels reported in the literature (60-110 micromol/L for adults males, 45-90 micromol/L for adult females) [10]. This criteria was chosen to align with the criteria used by the Fijian teaching hospital that is affiliated with the Fiji National University: the 200mcmol/L criteria reflects their AKI triage management guidelines based on the low-resourced context. The present study therefore adopted the same criteria to evaluate the similarly low-resourced context of Samoa. A total of 1185 patients were identified, and a request for their complete medical records was made to the Medical Record Department. Each record was reviewed for its suitability, and a total of 1071 records did not meet inclusion criteria. The sample size for the present study was therefore 114 patients.

The data collection form is an adaptation of the form used by the International Society for Nephrology for the Global Snapshot Project [11]. For each participant, the following information was collected:

2.2.1. Demographic and Baseline characteristics

* Demographic Information: age (years), gender (male/female), ethnicity (Samoan/Other).
* Admission Information: Admitting Department (Medica/Surgical/Obstetrics&Gynecology), risk factors for AKI (age>75 years/Diabetes Mellitus/Chronic Liver Disease/Chronic Heart Failure/Chronic Kidney Disease/anemia (Hb<9g/dL)/none/unknown), AKI acquisition (community/hospital), baseline serum creatinine within previous 12 months (micromole/L).
* Presenting symptoms for suspicion of AKI: Dehydration (diarrhea/vomiting/increased thirst/decreased intake), urinary symptoms (oliguria/polyuria/dysuria/heamaturia/incontinence/urolith passed), swelling (anasarca/face & neck/ upper limbs/ lower limbs/other), hypotension (MAP<65/shock and use of vasopressors/hemmorrhage), pregnancy and delivery-related symptoms (PV bleeding/coma/seizures/other), Fever, Traumatic injury (site), allergic reaction (specify), poisoning (specify).
* AKI KDIGO criteria-based diagnosis: increase in serum creatinine by 0.3 mg/dL or more within 48 hours OR, increase in serum creatinine to 1.5 times baseline or more within the last 7 days OR, urine output less than 0.5 mL/kg/h for 6 hours.

2.2.2. Aetiology

* Factors contributing to development of AKI: dehydration (diarrhea/vomiting/polyuria/decreased intake), liver (hepatorenal syndrome/cirrhosis/acute liver failure), cardiac (acute myocardial infarct/VHD/heart failure/pulmonary embolism/infective endocarditis/cardiorenal syndrome), hypotension and shock (cardiogenic shock/hemorrhage/sepsis/drug induced/anaphylaxis/post partum/hypotension of unclear cause), acute kidney diseases (acute glomerulonephritis/interstitial nephritis/pyelonephritis/rhabdomyolysis/intravascular hemolysis), urinary obstruction (sone/tumor/prostate condition), infections (leptospirosis/dengue/TB, other bacterial/other viral), pregnancy related (miscarriage with septic shock/puerperal sepsis), systemic diseases (multiple myeloma/SLE/DIC/pre-eclampsia/PPH/hyperemesis gravidarum), nephrotoxic agents (ACEI/ARB, NSAIDS, aminoglycosides/chemotherapy/contrast), poisoning (yes/no).
* Blood parameter on the day AKI was confirmed: Urea (umol/L), creatinine (umol/L), urine output in past 24 hours (mls).
* Known infection site (yes/no), and if yes specify infection site.
* Other organ failures: pulmonary, cardiovascular, hepatic, hematological, neurological, none.

2.2.3. Management

* Non-dialytic treatment at the time of AKI diagnosis: fluid therapy, diuretics, vasosupressors, antibiotics, urinary diversion (percutaneous nephrostomy, cystectomy, urethral catheterization), fluid restriction, other.
* Patient received dialysis (yes/no).
* Indication for starting dialysis: fluid overload, symptomatic uremia, electrolyte or acid-based disturbance, intoxication/poisoning, other.
* Number of days from diagnosis of AKI to initiation of haemodialysis (days).
* Blood parameters on the day hemodialysis was started: Urea (umol/L), creatinine (umol/L), urine output in past 24 hours (mls).

2.2.4. Outcome

* Patient status: Alive/deceased.
* Cause of death: kidney failure, infection/sepsis, cardiovascular, shock, dehydration, hemorrhage, pregnancy-related, liver failure, pulmonary condition, neurological, trauma, poisoning, systemic illness, malignancy, unknown.

2.3. Data analysis The data was analysed using the Microsoft Excel and STATA statistical software packages. Descriptive analysis and pivot tables were performed initially, followed by comparison of binary variables (unpaired t-test significant at p<0.05) and the unadjusted Kaplan Meier curve.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18 years) admitted to general wards of Tupua Tamasese Meaole (TTM) Hospital with a diagnosis of AKI between the 1st December 2019 and the 31st of May 2020
* serum creatinine level of >200 micromol/L
* compliance with the current Kidney Disease Improving Global Outcomes (KDIGO) criteria for AKI diagnosis

Exclusion Criteria:

* patients on chronic haemodialysis
* patients with underlying chronic kidney disease with no evidence of AKI
* patients for whom it was not possible to ascertain a diagnosis (i.e., patients with one elevated serum creatinine result and no subsequent follow-up haematology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to TTM Hospital in Samoa during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
aetiology of AKI | 6 months
  the causes of AKI will be retrieved from the medical records and tallied for reporting in group summary format
management options chosen to treat AKI | 6 months
  the management options chosen to treat AKI will be retrieved from the medical records and tallied for reporting in group summary format.
outcome of AKI cases presenting to the emergency department | 6 months
  the outcomes of AKI cases presenting to the emergency department will be retrieved from the medical records and tallied for reporting in group summary format

CONTACTS AND LOCATIONS:
Locations (1):
- Tupua Tamasese Meaole Hospital, Apia, QLD, Samoa

IPD SHARING:
Plan to Share IPD: No
At this time, there is no IPD plan.